CLINICAL TRIAL: NCT01296581
Title: Phase I, First in Human, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of X-82 in Patients With Advanced Solid Tumors
Brief Title: Safety Study of X-82 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tyrogenex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X82-CLI-101
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Advanced Solid Tumors
Keywords: Cancer; Tumors; VEGFR; PDGFR
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- X-82 (Experimental)
  Interventions: Drug: X-82

INTERVENTIONS:
Drug: X-82 — Dose escalation starting at 20 mg, oral once or twice a day, 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of X-82 as a single agent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced solid tumor malignancy that is not responsive to standard therapies or for which there is no effective therapy.
* Expansion Cohort Phase: Histologically or cytologically confirmed recurrent serous or clear cell epithelial ovarian adenocarcinoma, fallopian tube carcinoma, or primary peritoneal carcinoma for which there is no available curative standard therapy, in the investigator's opinion.
* Eastern Cooperative Group (ECOG) Performance Status score of 0 or 1.
* Life expectancy of at least 12 weeks.
* Ability to swallow and retain oral medication.
* Adequate organ system function.
* Male patients willing to use adequate contraceptive measures.
* Female patients who are not of child-bearing potential, and female patients of child-bearing potential who agree to use adequate contraceptive measures and who have a negative serum or urine pregnancy test within 24 hours prior to initial trial treatment.
* Patients must have measurable or evaluable disease.
* Expansion Cohort Phase: Patients with serous histology must have a CA 125 level ≥ 2x ULN within 14 days prior to the start of X-82. Patients with elevated CA 125 levels at baseline are not required to have measurable disease by RECIST criteria. Patients with clear cell histology that do not have an elevated CA 125 level must have measurable disease.
* Patients must be ≥ 18 years of age.
* Patients entering this study must be willing to provide tissue from a previous tumor biopsy (if available) for correlative testing. If tissue is not available, a patient will still be eligible for enrollment into the study. For the expansion cohort, patients will also be requested, but not required, to undergo a pre-treatment biopsy.
* Willingness and ability to comply with trial and follow-up procedures.
* Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

* Patients currently receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy [with the exception of LHRH agonists for prostate cancer], surgery and/or tumor embolization).
* Use of an investigational drug within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of X-82. A minimum of 10 days between termination of the investigational drug and administration of X-82 is required. In addition, any drug-related toxicity should have recovered to grade 1 or less.
* Any major surgery, radiotherapy, or immunotherapy within the last 21 days (limited palliative radiation is allowed ≥2 weeks). Chemotherapy regimens with delayed toxicity within the last 4 weeks (or within the last 6 weeks for prior nitrosourea or mitomycin C). Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last 2 weeks.
* Patients with a known allergy or delayed hypersensitivity reaction to drugs chemically related to X-82 (sunitinib, sorafenib or pazopanib) or to the active ingredient of X-82.
* Concomitant use of drugs with a risk of causing prolonged QTc and/or Torsades de Pointes.
* Concomitant use of herbal medications (i.e. St. John's wort, Kava, ephedra (ma huang), ginko biloba) at least 7 days prior to the first dose of study drug and throughout participation in the trial.
* Patients with known CNS metastases, unless metastases are treated and stable and the patients do not require systemic steroids
* Treatment with therapeutic doses of coumarin-type anticoagulants (maximum daily dose of 1mg allowed for port line patency permitted). Low molecular weight heparin (LMWH) will be allowed.
* Females who are pregnant or breastfeeding.
* Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of X-82.
* Decreased left ventricular function at study entry defined as LVEF <50% by either Echocardiogram or MUGA scan.
* Patients who have previously experienced myocardial infarction, severe/unstable angina, coronary/peripheral arterial bypass, symptomatic congestive heart failure (New York Heart Association [NYHA] Class 3 or 4), arterial thrombosis, cerebrovascular accident, or transient ischemia, in the 60 days prior to Day 1 of Cycle 1.
* Patients with inadequately controlled hypertension (defined as BP > 150/100) with or without current antihypertensive medications. Patients with a history of additional risk factors for Torsades de Pointes (e.g. familial long QT syndrome, heart failure, left ventricular hypertrophy, slow heart rate (<45 bpm).
* Patient with a QTcF interval ≥450 msecs or other significant ECG abnormalities as determined the investigator.
* A serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol
* Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol
* Patients with a history of intolerance to, or significant toxicity with, VEGFR tyrosine kinase inhibitor(s) (TKI).
* Patients entering the expansion after the determination of MTD are limited to previous treatment with one anti-VEGFR TKI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-02; Primary Completion 2014-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 12 months
  To determine the maximum tolerated dose (MTD) of X-82 as a single agent.

SECONDARY OUTCOMES:
Preliminary Pharmacokinetics of X-82 given as a single agent | 12 months
  To characterize the preliminary pharmacokinetics (PK) of X-82 given as a single agent.
Preliminary biological activity | 18 months
  To explore the preliminary biological activity and clinical tumor response after treatment with X-82 given as a single agent.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Courtney, MD, Principal Investigator — Study PI
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Bendell JC, Patel MR, Moore KN, Chua CC, Arkenau HT, Dukart G, Harrow K, Liang C. Phase I, First-in-Human, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Vorolanib in Patients with Advanced Solid Tumors. Oncologist. 2019 Apr;24(4):455-e121. doi: 10.1634/theoncologist.2018-0740. Epub 2018 Nov 26. PMID 30478190